CLINICAL TRIAL: NCT04815967
Title: Phase 2/3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Single-Treatment Efficacy and Safety Study of MYOBLOC in Treatment of Adult Upper Limb Spasticity and Open-Label Extension, Multiple-Treatment Safety Study of MYOBLOC
Brief Title: Efficacy and Safety Study of MYOBLOC® in the Treatment of Adult Upper Limb Spasticity
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Collaborators: Solstice Neurosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SN-SPAS-201
Record Dates: First submitted 2021-02-11; First posted 2021-03-25 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Spasticity; Cerebrovascular Accident; Multiple Sclerosis; Traumatic Brain Injury; Cervical Spinal Cord Injury; Cerebral Palsy
Keywords: Stroke; Traumatic Brain Injury; Monoplegia; Hemiplegia; Upper limb; Multiple Sclerosis; Cerebral Palsy; Cervical Spinal Cord Injury
MeSH Terms: conditions — Muscle Spasticity; Stroke; Multiple Sclerosis; Brain Injuries, Traumatic; Cerebral Palsy; Hemiplegia | interventions — Clinical Trials, Phase II as Topic; rimabotulinumtoxinB; Clinical Trials, Phase III as Topic

STUDY DESIGN:
Intervention Model Description: A Phase 2/3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Single-Treatment Efficacy and Safety Study of MYOBLOC in the Treatment of Adult Upper Limb Spasticity Followed by an Open-Label Extension, Multiple-Treatment in Safety Study of MYOBLOC
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No other parties are masked in the clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Phase 2; Low Dose MYOBLOC (Experimental): Low Dose MYOBLOC is a single treatment and will be compared to volume-matched placebo
  Interventions: Drug: Phase 2; Low Dose MYOBLOC
- Phase 2; High Dose MYOBLOC (Experimental): High Dose MYOBLOC is a single treatment and will be compared to volume-matched placebo
  Interventions: Drug: Phase 2; High Dose MYOBLOC
- Phase 2; Placebo (Placebo Comparator): Volume-matched placebo is a single treatment
  Interventions: Drug: Phase 2; Placebo
- Phase 3; MYOBLOC (Experimental): MYOBLOC is a single treatment and will be compared to volume-matched placebo
  Interventions: Drug: Phase 3; MYOBLOC
- Phase 3; Placebo (Placebo Comparator): Volume-matched placebo is a single treatment
  Interventions: Drug: Phase 3; Placebo

INTERVENTIONS:
Drug: Phase 2; Low Dose MYOBLOC — Intramuscular injections on Day 1
  Other Names: rimabotulinumtoxinB; botulinum toxin type B
  Arms: Phase 2; Low Dose MYOBLOC
Drug: Phase 2; High Dose MYOBLOC — Intramuscular injections on Day 1
  Other Names: rimabotulinumtoxinB; botulinum toxin type B
  Arms: Phase 2; High Dose MYOBLOC
Drug: Phase 2; Placebo — Intramuscular injections on Day 1
  Other Names: PBO
  Arms: Phase 2; Placebo
Drug: Phase 3; MYOBLOC — Intramuscular injections on Day 1
  Other Names: rimabotulinumtoxinB; botulinum toxin type B
  Arms: Phase 3; MYOBLOC
Drug: Phase 3; Placebo — Intramuscular injections on Day 1
  Other Names: PBO
  Arms: Phase 3; Placebo

SUMMARY:
Phase 2/3, randomized, double-blind, placebo-controlled, single-treatment, multicenter trial assessing the efficacy and safety of MYOBLOC for the treatment of upper limb spasticity in adults followed by an open-label extension safety trial.

DETAILED DESCRIPTION:
Phase 2, randomized, double-blind, placebo-controlled, single-treatment, multicenter trial will compare the efficacy and safety of two doses of MYOBLOC versus volume-matched placebo in the treatment of upper limb spasticity in adults. An interim analysis will evaluate all available safety and efficacy data from the Phase 2 double-blind trial in order to recommend which dose will be evaluated in subsequent Phase 3 trial. The Phase 3, randomized, double-blind, placebo-controlled, single-treatment, multicenter trial will compare the efficacy and safety of MYOBLOC versus placebo in the treatment of upper limb spasticity in adults. Subjects who complete either the Phase 2 or Phase 3 trial will continue into an open-label extension where each will receive 5 separate MYOBLOC treatments (~13 week apart) for upper limb spasticity.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Able to understand the potential risks and benefits, the study requirements, and provide written informed consent before enrollment into the study; or if unable, the subject's Legally Authorized Representative (LAR) may provide written informed consent.
2. Male or female ≥18 to maximum of 80 years of age, inclusive.
3. Upper limb spasticity due to stroke, or traumatic brain injury, or spinal cord injury that occurred ≥ 6 months prior to randomization. Eligible subjects may have upper limb monoplegia or hemiplegia. Subjects with cerebral palsy are eligible for study enrollment.
4. Modified Ashworth Scale (MAS) scores of ≥2 in at least two muscle groups inclusive of the elbow, wrist, and finger flexors at screening and baseline.
5. In the Investigator's opinion, the subject will be available and able to comply with the study requirements for at least 1 year, based on the subject's overall health and disease prognosis.
6. In the Investigator's opinion, the subject will be willing and able to comply with all requirements of the protocol, including completion of study questionnaires. A caregiver may be designated to assist with the physical completion of questionnaires/scales.

EXCLUSION CRITERIA:

1. Quadriplegia/tetraplegia, or triplegia with both upper limbs affected.
2. Uncontrolled epilepsy or any type of seizure disorder with a seizure(s) within the previous year.
3. Neuromuscular disorders including, but not limited to, amyotrophic lateral sclerosis (ALS), primary lateral sclerosis (PLS), multiple sclerosis (MS), myasthenia gravis, or muscular dystrophy.
4. History of major joint contracture(s), in which, based on the Investigator's assessment, the contracture(s) significantly contributes to joint immobility in the affected upper limb.
5. Unresolved fracture(s) in the affected upper limb.
6. Severe atrophy in the affected upper limb.
7. Known hypersensitivity to botulinum toxins type A or B or to any MYOBLOC solution components.
8. Concomitant use or exposure within 5 half-lives of randomization of the following: aminoglycoside antibiotics, curare-like agents, or other agents that may interfere with neuromuscular function.
9. Treatment with a neurolytic agent (e.g., phenol, alcohol blocks) to the affected upper limb within 1 year before randomization.
10. Presence of a spinal stimulator or intrathecal baclofen pump that has not been turned off within 30 days prior to screening.
11. Changes to treatment regimen or any new treatment with oral antispasmodics and/or muscle relaxants within 30 days prior to randomization.
12. Initiation of physical and/or occupational therapy <30 days before randomization. Subjects receiving physical and/or occupational therapy ≥30 days before randomization must be willing to maintain their therapy regimen through Week 4 of the Double-Blind Period.
13. Prior botulinum toxin type A (BoNT/A) or B (BoNT/B) treatment in the affected upper limb within 24 weeks before screening. Prior BoNT/A or BoNT/B treatment in areas other than the affected upper limb is not exclusionary but must have occurred at least 12 weeks before screening. Prior toxin exposure must have been well tolerated and without any significant long-term side effects in the case of repeated prior exposure.
14. Subjects should not receive nor have any plans to receive any botulinum toxin treatment, other than the study drug (MYOBLOC), from the time that informed consent is obtained until participation in the study is complete.
15. Severe dysphagia (i.e., inability to swallow liquids, solids or both without choking or medical intervention), or dysphagia with a history of aspiration pneumonia, within 6 months before screening.
16. Prior surgery to treat spasticity in the affected upper limb (i.e., tendon lengthening or tendon transfer).
17. Any anticipated or scheduled surgery during the study period, with the exception of dermatological procedures performed under local anesthesia for the purposes of removing precancerous and cancerous lesions.
18. Major surgery within 30 days before screening.
19. Pregnancy or breastfeeding.
20. Females of childbearing potential must agree to practice a medically acceptable method of contraception (e.g., intrauterine device, hormonal contraception started at least one full cycle before study enrollment, or barrier method in conjunction with spermicide) for the duration of the study (including 2 months after study completion). For the purposes of this study, all females are considered to be of childbearing potential unless they are confirmed by the Investigator to be post-menopausal (at least 1 year since last menses and laboratory test confirmation), biologically sterile, or surgically sterile (e.g., hysterectomy with bilateral oophorectomy, tubal ligation).
21. History of drug or alcohol abuse within 6 months before screening.
22. Obstructive pulmonary disease with forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) <70%.
23. Slow vital capacity (SVC) <60% of predicted.
24. Chronic or current use of inhaled corticosteroids.
25. Ventilator dependence (i.e., 24-hour ventilator dependence when intubated, or due to a failure to wean the subject from the ventilator while hospitalized in the intensive care unit or respiratory care center). Subjects who use oxygen on an as-needed basis or during sleeping hours only via a nasal cannula are eligible for the study.
26. Infection at the planned sites of injection.
27. Treatment with an investigational drug, device, or biological agent within 30 days before screening or while participating in this study.
28. Malignancy diagnosed 3 months before screening.
29. Has one or more screening clinical laboratory test values outside the reference range that, in the opinion of the Investigator, are clinically significant, or any of the following :

    * Serum creatinine >1.5 times the upper limit of normal (ULN);
    * Serum total bilirubin > 1.5 times ULN;
    * Serum alanine aminotransferase or aspartate aminotransferase >2 times ULN.
30. Has any of the following cardiac findings at screening:

    * Abnormal ECG that is, in the Investigator's opinion/evaluation, clinically significant;
    * PR interval >220 ms;
    * QRS interval >130 ms;
    * QTcF interval >450 ms (for men), or >470 ms (for women) (QT corrected using Fridericia's method);
    * Second-or third-degree atrioventricular block;
    * Any rhythm, other than sinus rhythm, that is interpreted or assessed by the Investigator to be clinically significant.
31. Any other medical illness, condition, or clinical finding that, in the opinion of the Investigator and/or the Sponsor, would put the subject at undue risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Effect of MYOBLOC on the Modified Ashworth Scale (MAS) for tone of the Primary Target Muscle Group (PTMG) [Phase 2 and Phase 3] | Baseline and Week 4
  The first co-primary endpoint is the change from baseline in Modified Ashworth Scale (MAS) score for tone of the Primary Target Muscle Group (PTMG) selected for treatment at Week 4 post-injection. The MAS is an internationally accepted and validated instrument used to measure resistance during passive soft-tissue stretching. Resistance will be measured and recorded using a 6-point scale ranging from 0 (no increase in muscle tone) to 4 (affected part[s] rigid in flexion or extension). A lower change from baseline MAS score (<0) represents a better outcome.
Effect of MYOBLOC on Clinical Global Impression of Change (CGI-C) Scale [Phase 2 and Phase 3] | Week 4
  The second co-primary endpoint is the Clinical Global Impression of Change (CGI-C) score in functional ability at Week 4 post-injection. The CGI-C scale is a single item clinician assessment of how much the patient's functional ability has improved, worsened or has not changed relative to the patient's baseline state prior to treatment (injection). The CGI-C is rated on a 7-point Likert scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". Successful therapy is indicated by a lower score (<4) in subsequent testing.

SECONDARY OUTCOMES:
Effect of MYOBLOC on the Modified Ashworth Scale (MAS) for tone in each muscle group selected for treatment [Phase 2 and Phase 3] | Baseline and Week 4
  An additional secondary endpoint is the change from baseline in Modified Ashworth Scale (MAS) score for tone in each muscle group selected for treatment at Week 4 post-injection. The MAS is an internationally accepted and validated instrument used to measure resistance during passive soft-tissue stretching. Resistance will be measured and recorded using a 6-point scale ranging from 0 (no increase in muscle tone) to 4 (affected part[s] rigid in flexion or extension). A lower change from baseline MAS score (<0) represents a better outcome.
Effect of MYOBLOC on the Patient Global Impression of Change (PGI-C) [Phase 2 and Phase 3] | Week 4
  An additional secondary endpoint is the Patient Global Impression of Change (PGI-C) score at Week 4 post-injection. The PGI-C scale is a single item patient reported (self) assessment of how much his/her ability to function has improved, worsened or has not changed relative to his/her baseline state prior to treatment (injection). The PGI-C is rated on a 7-point Likert scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". Successful therapy is indicated by a lower score (<4) in subsequent testing.
Effect of MYOBLOC on the Caregiver Global Impression of Change (GGI-C) [Phase 2 and Phase 3] | Week 4
  An additional secondary endpoint is the Caregiver Global Impression of Change (GGI-C) score at Week 4 post-injection. The GGI-C scale is a single item caregiver assessment on how much the patient's ability to function has improved, worsened or has not changed relative to the patient's baseline state prior to treatment (injection). The GGI-C is rated on a 7-point Likert scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". Successful therapy is indicated by a lower score (<4) in subsequent testing.
Effect of MYOBLOC on the Pain Numeric Rating Scale (Pain-NRS) [Phase 2 and Phase 3] | Baseline and Week 4
  An additional secondary endpoint is the change from baseline in the Pain Numeric Rating Scale (Pain-NRS) score at Week 4 post-injection. The Pain-NRS is a unidimensional measure of pain intensity in adults. It is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. Similar to the VAS, the Pain-NRS is anchored by terms describing pain severity on 11-point scale ranging from 0 ("no pain") to 10 ("worse pain imaginable"). A lower change from baseline Pain-NRS score (<0) represents a better outcome.
Effect of MYOBLOC on the Modified Barthel Index (MBI) [Phase 2 and Phase 3] | Baseline and Week 4
  An additional secondary endpoint is the change from baseline in the Modified Barthel Index (MBI) score at Week 4 post-injection. The MBI is a 10-item self-assessment scale that measures the patient's degree of independence with activities of daily living (bowel control, bladder control, help with grooming, toilet use, feeding, transfers, walking, dressing, climbing stairs, and bathing). An item (activity) is given one of five levels (ratings) of dependency ranging from 0 (unable to perform task) to a maximum of 5, 10, or 15 (fully independent). The sum of ratings of the 10 items yields a total score ranging from 0 to 100. A higher change from baseline MBI score (>0) represents a better outcome.
Effect of MYOBLOC on the Modified Ashworth Scale (MAS) Responder Rate for the Primary Target Muscle Group (PTMG) [Phase 2 and Phase 3] | Baseline and Week 4
  An additional secondary endpoint is the Modified Ashworth Scale (MAS) Responder Rate for the Primary Target Muscle Group (PTMG) at Week 4 post-injection. The MAS responder rate is defined as the percent of subjects with ≥1 grade reduction in their change from baseline MAS score for the PTMG at Week 4. Values range from 0 to 100%. A higher percentage represents a greater number of responders.
Effect of MYOBLOC on the Modified Ashworth Scale (MAS) for tone in the Primary Target Muscle Group (PTMG) [Phase 2 and Phase 3] | Baseline and Weeks 2, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary endpoint is the change from baseline in Modified Ashworth Scale (MAS) score for tone in the Primary Target Muscle Group (PTMG) at Weeks 2, 8 and 13 (and, if applicable, at re-evaluation visit) post-injection. The MAS is an internationally accepted and validated instrument used to measure resistance during passive soft-tissue stretching. Resistance will be measured and recorded using a 6-point scale ranging from 0 (no increase in muscle tone) to 4 (affected part[s] rigid in flexion or extension). A lower change from baseline MAS score (<0) represents a better outcome.
Effect of MYOBLOC on the Modified Ashworth Scale (MAS) for tone in each muscle group selected for treatment [Phase 2 and Phase 3] | Baseline and Weeks 2, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary endpoint is the change from baseline in Modified Ashworth Scale (MAS) score for tone in each muscle group selected for treatment at Weeks 2, 8 and 13 (and, if applicable, at re-evaluation visit) post-injection. The MAS is an internationally accepted and validated instrument used to measure resistance during passive soft-tissue stretching. Resistance will be measured and recorded using a 6-point scale ranging from 0 (no increase in muscle tone) to 4 (affected part[s] rigid in flexion or extension). A lower change from baseline MAS score (<0) represents a better outcome.
Effect of MYOBLOC on Clinical Global Impression of Change (CGI-C) Scale [Phase 2 and Phase 3] | Weeks 2, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary endpoint is the Clinical Global Impression of Change (CGI-C) score in functional ability at Weeks 2, 8, and 13 (and, if applicable, at re-evaluation visit) post-injection. The CGI-C scale is a single item clinician assessment of how much the patient's functional ability has improved, worsened or has not changed relative to the patient's baseline state prior to treatment (injection). The CGI-C is rated on a 7-point Likert scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". Successful therapy is indicated by a lower score (<4) in subsequent testing.
Effect of MYOBLOC on the Clinical Global Impression of Severity (CGI-S) [Phase 2 and Phase 3] | Baseline and Weeks 2, 4, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary efficacy endpoint is the change from baseline in the Clinical Global Impression of Severity (CGI-S) score at Weeks 2, 4, 8 and 13 (and, if applicable, at re-evaluation visit) post-injection. The CGI-S is a single item clinician assessment of the severity of impairment the patient's spasticity has on his or her ability to function based on the clinician's total clinical experience with patients with upper limb spasticity. The CGI-S is rated on a 7-point Likert scale from 1 to 7, where 1=normal; 2=borderline impaired; 3=mildly impaired; 4=moderately impaired; 5=markedly impaired; 6=severely impaired; 7=among the most extremely impaired. A change from baseline CGI-S score <0 represents a better outcome.
Effect of MYOBLOC on the Patient Global Impression of Change (PGI-C) [Phase 2 and Phase 3] | Weeks 2, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary endpoint is the Patient Global Impression of Change (PGI-C) score at Weeks 2, 8 and 13 (and, if applicable, at re-evaluation visit) post-injection. The PGI-C scale is a single item patient reported (self) assessment of how much his/her ability to function has improved, worsened or has not changed relative to his/her baseline state prior to treatment (injection). The PGI-C is rated on a 7-point Likert scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". Successful therapy is indicated by a lower score (<4) in subsequent testing.
Effect of MYOBLOC on the Patient Global Impression of Severity (PGI-S) [Phase 2 and Phase 3] | Baseline and Weeks 2, 4, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary efficacy endpoint is the change from baseline in the Patient Global Impression of Severity (PGI-S) score at Weeks 2, 4, 8, and 13 (and, if applicable, at re-evaluation visit) post-injection. The PGI-S is a single item patient reported (self) assessment of his/her severity of impairment their spasticity has on his or her ability to function. The PGI-S is rated on a 7-point Likert scale from 1 to 7, where 1=normal; 2=borderline impaired; 3=mildly impaired; 4=moderately impaired; 5=markedly impaired; 6=severely impaired; 7=among the most extremely impaired. A change from baseline PGI-S score <0 represents a better outcome.
Effect of MYOBLOC on the Caregiver Global Impression of Change (GGI-C) [Phase 2 and Phase 3] | Weeks 2, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary endpoint is the Caregiver Global Impression of Change (GGI-C) score at Weeks 2, 8 and 13 (and, if applicable, at re-evaluation visit) post-injection. The GGI-C scale is a single item caregiver assessment on how much the patient's ability to function has improved, worsened or has not changed relative to the patient's baseline state prior to treatment (injection). The GGI-C is rated on a 7-point Likert scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". Successful therapy is indicated by a lower score (<4) in subsequent testing.
Effect of MYOBLOC on the Caregiver Global Impression of Severity (GGI-S) [Phase 2 and Phase 3] | Baseline and Weeks 2, 4, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary efficacy endpoint is the change from baseline in the Caregiver Global Impression of Severity (GGI-S) score at Weeks 2, 4, 8 and 13 (and, if applicable, at re-evaluation visit) post-injection. The GGI-S is a single item caregiver assessment of the severity of impairment the patient's spasticity has on his or her ability to function. The GGI-S is rated on a 7-point Likert scale from 1 to 7, where 1=normal; 2=borderline impaired; 3=mildly impaired; 4=moderately impaired; 5=markedly impaired; 6=severely impaired; 7=among the most extremely impaired. A change from baseline GGI-S score <0 represents a better outcome.
Effect of MYOBLOC on the Pain Numeric Rating Scale (Pain-NRS) [Phase 2 and Phase 3] | Baseline and Weeks 2, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary endpoint is the change from baseline in the Pain Numeric Rating Scale (Pain-NRS) score at Weeks 2, 8 and 13 (and, if applicable, at re-evaluation visit) post-injection. The Pain-NRS is a unidimensional measure of pain intensity in adults. It is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. Similar to the VAS, the Pain-NRS is anchored by terms describing pain severity extreme on 11-point scale ranging from 0 ("no pain") to 10 ("worse pain imaginable"). A lower change from baseline Pain-NRS score (<0) represents a better outcome.
Effect of MYOBLOC on the Modified Barthel Index (MBI) [Phase 2 and Phase 3] | Baseline and Weeks 2, 8, and 13 (and, if applicable, at re-evaluation visit)
  An additional secondary endpoint is the change from baseline in the Modified Barthel Index (MBI) score at Weeks 2, 8 and 13 (and, if applicable, at re-evaluation visit) post-injection. The MBI is a 10-item scale self assessment that measures the patient's degree of independence with activities of daily living (bowel control, bladder control, help with grooming, toilet use, feeding, transfers, walking, dressing, climbing stairs, and bathing). An item (activity) is given one of five levels (rating) of dependency ranging from 0 (unable to perform task) to a maximum of 5, 10, or 15 (fully independent). The sum of ratings of the 10 items yields a total score ranging from 0 to 100. A higher change from baseline MBI score (>0) represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, MD, MBA, Study Chair — Supernus Pharmaceuticals
Locations (9):
- United States (7):
  - Rancho Research Institute, Downey, California
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Idaho Physical Medicine and Rehabilitation, Boise, Idaho
  - Coastal Neurology, Port Royal, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Czechia (2):
  - Fakultní nemocnice Brno, Neurologická klinika FN Brno (University Hospital Brno, Department of Neurology), Brno
  - Centrum pro intervenční terapii motorických poruch, Neurologická klinika, Univerzita Karlova Katerinska, Prague

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.